CLINICAL TRIAL: NCT02122718
Title: Xanthine Oxidase Inhibition for Improvement of Long-term Outcomes Following Ischaemic Stroke and Transient Ischaemic Attack
Brief Title: XILO-FIST, the Effect of Allopurinol on the Brain Heart and Blood Pressure After Stroke
Acronym: XILO-FIST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GN12MT494; TSA BHF 2013/01 (Other Grant/Funding Number: The Stroke Association)
Record Dates: First submitted 2014-04-23; First posted 2014-04-24 (Estimated); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Ischaemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol (Experimental)
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol
  Arms: Allopurinol
Drug: Placebo
  Arms: Placebo

SUMMARY:
Recurrent stroke and cognitive decline are common after ischaemic stroke. Allopurinol, a drug usually used to treat gout, has been shown to reduce heart ischaemia, heart size, and arterial stiffness and to relax brain blood vessels and may reduce the blood pressure. All of these properties may be associated with a lower risk of second stroke and cognitive decline. We now aim to explore whether allopurinol will reduce further damage to the brain (called white matter hyper-intensities) after stroke and also whether it reduces heart size and blood pressure after stroke.

We will conduct a multi-centre randomised, double-blind placebo controlled study to investigate whether two years allopurinol 300 mg twice per day (BD) improves these 3 outcomes, which are inextricably linked to risk of recurrence and cognitive decline after ischaemic stroke.

DETAILED DESCRIPTION:
New strategies are needed to improve long-term outcomes after ischaemic stroke or transient ischaemic attack (TIA). Approximately 13% of participants suffered recurrent stroke in recent secondary preventative trials , 40% of patients with TIA experience recurrent cardiovascular (CV) events during long-term follow up and there is an additional substantial burden from incident post-stroke dementia (~ 10% after first stroke and higher still after recurrent events) , cognitive decline (over 30%) and decline in physical function. Improving these outcomes is a recognised priority area for stroke research (as identified by stroke survivors through the recent James Lind Alliance priority setting workshops ).

Such adverse outcomes are particularly common in those with brain white matter hyper-intensities (WMH) on brain magnetic resonance imaging (MRI) . WMH are seen in as many as 90% of patients with ischaemic stroke , , are at least moderately severe in 50%6 and such 'severe' WMH are associated with substantially higher stroke recurrence rates (43% in one study)6, death and increased cognitive and physical decline. The burden of WMH increases during longitudinal follow up and this is associated with increased incident stroke, dementia and cognitive decline5. In the longitudinal population based Rotterdam scan study, 39% of elderly participants had WMH progression (over a mean period of 3.4 years) , as did 50% in the recent PROFeSS MRI sub-study (over 2 years)7 and 74% (over 3 years) in the Leukoariosis and Disability study (LADIS) .Similarly, silent brain infarction (SBI) is also associated with recurrent stroke and 14% developed incident infarcts on brain MRI in the Rotterdam scan study9. Thus, treatments that reduce WMH progression and incident silent brain infarction could have potentially profound effects on a variety of outcomes after stroke including cognition, functional outcome and recurrent stroke.

The pathological basis for WMH development and progression is poorly understood. Post mortem studies show presence of varied pathologies including demyelination, infarction, arteriosclerosis and breakdown of the blood-brain barrier. Key risk factors for development and progression of WMH are age, arterial hypertension and previous stroke9 and associations with other cardiovascular risk factors and left ventricular hypertrophy (LVH) have been demonstrated . Blood pressure (BP) lowering reduces WMH progression, as demonstrated by the PROGRESS MRI sub-study . In the PROFeSS MRI sub-study WMH progression was unaffected by the angiotensin receptor blocker telmisartan7 but unlike PROGRESS, there was no significant difference in BP between groups. In addition, WMH are less clearly related to hypertension in older patients with established cardiovascular disease meaning that novel strategies which reduce WMH progression and SBI would be particularly promising in this group.

The association between WMH and LVH is of particular interest; it appears independent of arterial BP , and may be mediated by aortic stiffness . There are additional potential mechanisms for this association (e.g., LVH is the strongest predictor of left atrial appendage thrombi, stronger than any left atrial parameter) . Regression of LVH is associated with reduced risk of stroke. In a recent meta-analysis of 14 studies in 12,809 patients, LVH regression was independently associated with a 25% reduction in future strokes, whereas the composite endpoint of CV events/mortality was only 15% lower . Similar findings were seen in the LIFE echo sub-study which utilised measures of left ventricular mass (LVM) . LVH regression is thus a promising therapeutic target in devising new ways to prevent strokes, especially if the same treatment were found to reduce WMH.

ELIGIBILITY:
Inclusion Criteria:

* Ischaemic Stroke/ Ischaemic lesion on brain imaging in relevant anatomical territory in patients with transient ischaemic attack.
* Age greater than 50 years. -- Consent within one month of stroke.

Exclusion Criteria:

* Modified Rankin scale score of 5 (at end of the possible enrolment window of one month after stroke).
* Diagnosis of dementia (defined as a documented diagnosis or a screening Informant Questionnaire for Cognitive Decline in the Elderly (IQCODE) score of 3.6 or more).
* Cognitive impairment deemed sufficient to compromise capacity to consent or to comply with the protocol (in the opinion of the local investigator).
* Dependent on daily help from others for basic or instrumental activities of daily living prior to stroke (defined as assistance needed with toileting, walking or dressing).
* Significant co-morbidity or frailty likely to cause death within 24 months or likely to make adherence to study protocol difficult for participant (in the opinion of the local investigator).
* Contra-indication to or indication for administration of allopurinol (as detailed in Summary of Product Characteristics on the XILO-FIST web portal and in trial master file).
* Concurrent azathioprine, 6-mercaptopurine therapy, other cytotoxic therapies, cyclosporin, theophylline and didanosine.
* Significant hepatic impairment (defined as serum bilirubin, Aspartate Aminotransferase (AST) or Alanine transaminase (ALT) greater than three times upper limit of normal (ULN)).
* Estimated Glomerular Filtration Rate < 30 mls/min
* Contraindication to MRI scanning.
* Women who are pregnant or breastfeeding.
* Women of childbearing potential who are unable or unwilling to use contraception.
* Prisoners.
* Active participation in another Clinical Trial of Investigational Medicinal Product (CTIMP) or device trial or participation within the past month.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2014-05; Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
White matter hyper-intensities (WMH) progression rate over 2 years, defined using the Rotterdam Progression Score | 2 years

SECONDARY OUTCOMES:
change in mean day-time systolic BP at 1 month | 1 month
change in mean day-time diastolic BP at 1 month | 1 month
Schmidt's Progression Score | 2 years
Fazekas score | 2 years
Scheltens scale score | 2 years
New brain infarction on MRI | 2 years
Rotterdam Progression Score with those who die / become too frail to undergo MRI being assigned the highest score | 2 years
Montreal Cognitive Assessment (MoCA) score | 2 years
Incident dementia | 2 years
change in mean day-time systolic BP at 2 years | 2 years
change in mean day-time diastolic BP at 2 years | 2 years
blood pressure variability | 2 years
Quality of life (EQ-5D, Stroke Specific Quality of Life Scale (SS-QOL)) | 2 years
Recurrent stroke | 2 years
Recurrent myocardial infarction (MI), stroke or cardiac death | 2 years
Mortality | 2 years
Incident atrial fibrillation | 2 years
Clinic blood pressure | 2 years

OTHER OUTCOMES:
Cardiac sub-study: Change in measured Left ventricular mass (LVM) at 2 years | 2 years
Cardiac sub-study: change in ejection fraction | 2 years
Cardiac Sub-study: change in end diastolic volume | 2 years
Cardiac sub-study: change in end systolic volume | 2 years
Cardiac Sub-study: change in stroke volume | 2 years
Cardiac sub-study: change in left atrial diameter | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Dawson, Principal Investigator — University of Glasgow
Locations (21):
- United Kingdom (21):
  - Altnagelvin Campus, Londonderry, County Derry
  - Broomfield Hospital, Chelmsford, Essex
  - Southend University Hospital, Westcliff-on-Sea, Essex
  - Darent Valley Hospital, Dartford, Kent
  - The Royal London Hospital, Whitechapel, London
  - Northumbria NHS Trust, Ashington, Northumberland
  - Royal United Hospital, Bath, Somerset
  - Royal Stoke University Hosptial, Stoke-on-Trent, Staffordshire
  - NHS Grampian, Aberdeen
  - NHS Lanarkshire, Airdrie
  - NHS Tayside, Dundee
  - South West Acute Hospital, Enniskillen
  - NHS Greater Glagsow and Clyde, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Barnet Hospital, London
  - Guys and St Thomas NHS Foundation Trust, London
  - UCL Stroke Research Centre, London
  - Luton and Dunstable University Hosptial, Luton
  - Newcastle UPon Tyne Hospitals NHS Trust, Newcastle
  - Nottingham University, Nottingham
  - City Hospital Sunderland NHS Foundation Trust, Sunderland

REFERENCES:
- [Derived] Dawson J, Robertson M, Dickie DA, Bath P, Forbes K, Quinn T, Broomfield NM, Dani K, Doney A, Houston G, Lees KR, Muir KW, Struthers A, Walters M, Barber M, Bhalla A, Cameron A, Dyker A, Guyler P, Hassan A, Kearney MT, Keegan B, Lakshmanan S, Macleod MJ, Randall M, Shaw L, Subramanian G, Werring D, McConnachie A. Xanthine oxidase inhibition and white matter hyperintensity progression following ischaemic stroke and transient ischaemic attack (XILO-FIST): a multicentre, double-blinded, randomised, placebo-controlled trial. EClinicalMedicine. 2023 Feb 16;57:101863. doi: 10.1016/j.eclinm.2023.101863. eCollection 2023 Mar. PMID 36864979
- [Derived] Dawson J, Broomfield N, Dani K, Dickie DA, Doney A, Forbes K, Houston G, Kean S, Lees K, McConnachie A, Muir KW, Quinn T, Struthers A, Walters M. Xanthine oxidase inhibition for the improvement of long-term outcomes following ischaemic stroke and transient ischaemic attack (XILO-FIST) - Protocol for a randomised double blind placebo-controlled clinical trial. Eur Stroke J. 2018 Sep;3(3):281-290. doi: 10.1177/2396987318771426. Epub 2018 Apr 18. PMID 30246149